CLINICAL TRIAL: NCT04519593
Title: ABSOLUTELY: A Multicenter Randomized Controlled Trial of Temporary Uterine Blood Supply Occlusion for Laparoscopic Myomectomy in Patients With UTErine LeiomYoma
Brief Title: ABSOLUTELY: A Temporary Uterine Blood Supply Occlusion for Laparoscopic Myomectomy in Patients With UTErine LeiomYoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mother and Child Clinic Saint-Petersburg (Other)
Responsible Party: Principal Investigator, Andrey Dubinin, MD, PhD, Gynecologist, Mother and Child Clinic Saint-Petersburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCCSPb-8-12-2020
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Uterine Leiomyoma; Uterine Fibroid; Leiomyoma, Uterine; Myoma;Uterus; Laparoscopic Myomectomy; Postoperative Complications; Blood Loss, Surgical; Fertility Issues; Pregnancy Complications
Keywords: temporary uterine artery occlusion; temporary uterine blood supply occlusion
MeSH Terms: conditions — Myofibroma; Leiomyoma; Postoperative Complications; Blood Loss, Surgical; Infertility; Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: Patients who meet study inclusion criteria will be randomized into one of two treatment arms: 1) laparoscopic myomectomy preceded by temporary uterine blood supply occlusion or 2) laparoscopic myomectomy with a conventional approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic myomectomy with temporary blood supply occlusion (Experimental): Laparoscopic myomectomy is performed with prior visualization and temporary bilateral clipping of uterine/internal iliac arteries and suspensory ligaments of ovaries.
  Interventions: Procedure: Laparoscopic myomectomy with prior temporary uterine blood supply occlusion
- Conventional laparoscopic myomectomy (Active Comparator): Laparoscopic myomectomy is performed without prior temporary blood supply occlusion.
  Interventions: Procedure: Conventional laparoscopic myomectomy

INTERVENTIONS:
Procedure: Laparoscopic myomectomy with prior temporary uterine blood supply occlusion — Visualization and temporary bilateral clipping of uterine/internal iliac arteries and suspensory ligaments of ovaries.
  Other Names: Temporary uterine arteries occlusion
  Arms: Laparoscopic myomectomy with temporary blood supply occlusion
Procedure: Conventional laparoscopic myomectomy — Laparoscopic myomectomy without prior temporary uterine blood supply occlusion
  Arms: Conventional laparoscopic myomectomy

SUMMARY:
A phase 3 multicenter unblinded randomized controlled trial comparing the temporary uterine blood supply occlusion with conventional approach during laparoscopic myomectomy in patients with uterine leiomyoma.

DETAILED DESCRIPTION:
Primary endpoints

• Assess the volume of blood loss

Secondary endpoints

* Compare the rates of intra- and postoperative complications, the necessity of blood transfusion, length of surgery, length of hospital and ICU stay, and leiomyoma symptoms relief
* Determine the procedure impact on fertility by evaluating the level of anti-mullerian hormone, pregnancy rates, pregnancy complications, and the way of delivery

Patients who meet study inclusion criteria will be randomized into one of two treatment arms: 1) laparoscopic myomectomy preceded by temporary uterine blood supply occlusion or 2) laparoscopic myomectomy with a conventional approach.

Sixty patients will undergo laparoscopic myomectomy preceded by temporary uterine blood supply occlusion performed by gynecologists at Mother and Child Clinic Saint-Petersburg and other institutions participating in the study. Sixty patients will undergo conventional laparoscopic myomectomy performed by gynecologists at Mother and Child Clinic Saint-Petersburg and other institutions participating in the study.

Patients eligible for inclusion, after signing an informed voluntary consent to participate in the study, will be randomized in a 1:1 ratio to the treatment groups using stratification by age, size, and leiomyoma nodes location.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic uterine leiomyoma
* Size of leiomyoma node >5 cm based on imaging
* Leiomyoma node types 3, 4, 5, 6 according to The International Federation of Gynecology and Obstetrics (FIGO) classification or type 2 not feasible to be removed during hysteroscopy
* Single or multiple nodes
* Absent contraindications for laparoscopic myomectomy
* Voluntarily signed informed consent to participate in the study

Exclusion Criteria:

* Age < 18 years
* Asymptomatic uterine leiomyoma
* Size of leiomyoma node <5 cm based on imaging
* Absence of leiomyoma node types 3, 4, 5, 6 according to FIGO classification and type 2 not feasible to be removed during hysteroscopy
* Planned simultaneous hysteroscopy with leiomyoma node excision
* Current pregnancy and breastfeeding
* Suspicion of a malignant uterine tumor
* Prior uterine leiomyoma surgery
* Contraindications for laparoscopic myomectomy
* Lack of decision-making capacity hindering signing the consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-27 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss | At the end of the intervention
  Evaluation of blood loss volume

SECONDARY OUTCOMES:
Treatment characteristics | During 6 months since the intervention
  Rates of intra- and postoperative complications, necessity of blood transfusion, length of surgery, length of hospital and ICU stay, leiomyoma symptoms relief
Impact on fertility | During 18 months since the intervention
  Level of anti-mullerian hormone, rate of pregnancy, pregnancy complications, the way of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Mother and Child Clinic Saint-Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No